CLINICAL TRIAL: NCT00717756
Title: Lenalidomide for Advanced Hepatocellular Cancer:A Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Memorial Hospital of Rhode Island (Other); Roger Williams Medical Center (Other)
Responsible Party: Principal Investigator, howard safran, Principle Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-HC-212; Celgene # RV-HCC-PI- 0159 (Other: brown university); celgene (Other: brown university)
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Liver Cancer
Keywords: liver cancer, second line
MeSH Terms: conditions — Liver Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — 25 mg po qd x 21 days then 1 week off equals one cycle
  Other Names: revlimid

SUMMARY:
This study will determine whether lenalidomide has activity in patients with advanced liver cancer that have had growth of their cancer after sorafenib.

DETAILED DESCRIPTION:
This study will determine the response rate and toxicities of lenalidomide as second line treatment for patients with liver cancer who have progressed after sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed HCC or triple phase CT consistent with HCC in a patient with known cirrhosis and AFP > 200 ng/ml.
2. Disease not amenable to curative surgical resection
3. Patients must have been previously treated with sorafenib. Patients who are unable to receive sorafenib due to financial reasons are also eligible.
4. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
5. No previous thalidomide.
6. Patients must have radiologically assessable tumor.
7. ECOG performance status of 0-2 at study entry.
8. Understand and voluntarily sign an informed consent form.
9. Age >18 years at the time of signing the informed consent form.
10. Able to adhere to the study visit schedule and other protocol requirements.
11. Laboratory test results within these ranges:

    * Absolute neutrophil count > 1000/mm3
    * Platelet count > 60,000/mm3
    * Serum creatinine > 2.0 mg/dL
    * Total bilirubin > 4 mg/dL
    * AST (SGOT) and ALT (SGPT) > 5 x ULN.
12. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix: H Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix: F Education and Counseling Guidance Document
13. Disease free of prior malignancies for > 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV. (The effect of immune modulation of lenalidomide on patients who are HIV positive is unknown).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Montefiore Medical Center, The Bronx, New York
  - Memorial Hospital of Rhode island, Pawtucket, Rhode Island
  - Lifespan Hospitals, Providence, Rhode Island

REFERENCES:
- [Result] Safran H, Charpentier KP, Kaubisch A, Mantripragada K, Dubel G, Perez K, Faricy-Anderson K, Miner T, Eng Y, Victor J, Plette A, Espat J, Bakalarski P, Wingate P, Berz D, Luppe D, Martel D, Rosati K, Aparo S. Lenalidomide for second-line treatment of advanced hepatocellular cancer: a Brown University oncology group phase II study. Am J Clin Oncol. 2015 Feb;38(1):1-4. doi: 10.1097/COC.0b013e3182868c66. PMID 23648434

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 60.5 [17 to 88]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 25
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by Recist Criteria
Description: radiographic response defined as partial response defined by RECIST:At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
  It is noted that while on average the time frame for scans was 4 months, there were two patients who at 32 and 36 months had not progressed.
Time Frame: on average about every 2 months until progression, on average about 4 months.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 40
participants | 6

ADVERSE EVENTS:
Time Frame: From time of signing consent to approximately 30 days post last dose of drug, for a maximum of 4 years
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=40)
edema gr 3, lethargy gr 2, HGB gr 2, hypotension gr 2 (Investigations) | 1 (1)
vasovagal episode gr3 (Investigations) | 1 (1)
ascites gr3, Liver dysfunction gr 3, fatigue gr 3, dehydration gr 3, vomiting gr 2, constipation gr2 (Investigations) | 1 (1)
bilirubin gr4, ascites gr 3, hyponatremia gr 3, hyperk gr 3 (Investigations) | 1 (1)
non-blistering rash gr 3 (Investigations) | 1 (1)
increased confusion (Investigations) | 1 (1)
muscle weakness gr3, myelosuppresion gr 3 (Investigations) | 1 (1)
bilirubin gr 3, right upper quad pain gr 2 (Investigations) | 1 (1)
n gr1, v gr1, d gr1, pain abd gr2, pain chest gr2, gastro viral gr2 (Investigations) | 1 (1)
fracture gr 2 (Investigations) | 1 (1)
syncope gr3 (Investigations) | 1 (1)
syncope gr3, enceph gr 5, liver failure gr 5, GI bleed gr 3, death gr 5 (Investigations) | 1 (1)
hepatic enceph gr 3, mood alteration gr 2, mental status change gr 3 (Investigations) | 1 (1)
lower chest pressure (Investigations) | 1 (1)
dizziness gr 3, dyspnea gr2, tumor pain gr 3, dehydration gr 3, confusion gr 1 (Investigations) | 1 (1)
bronchitis, pleural effusion, dyspnea, lower extrem edema, rash (Investigations) | 1 (1) — Labs AEs with SAE: anemia, ammonia, AST, alk phos, sodium, K, chloride, mg, co2, anion gap, albumin, BNP, ca, PLT
fever gr 2, chills gr 2, bilary obstruction gr2, sepsis gr 2 (Investigations) | 1 (1)
expired secondary to disease (Investigations) | 11 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=40)
alk phos (Investigations) | 4 (4)
alopecia (Investigations) | 3 (3)
ALT /AST (Investigations) | 7 (7)
ANC (Investigations) | 6 (6)
anemia (Investigations) | 6 (6)
anorexia (Investigations) | 4 (4)
ascites (Investigations) | 2 (2)
Ca (Investigations) | 3 (3)
constipation (Investigations) | 8 (8)
diarrhea (Investigations) | 5 (5)
diverticulitis (Investigations) | 2 (2)
dyspepsia (Investigations) | 3 (3)
edema (Investigations) | 4 (4)
esophageal stricture (Investigations) | 2 (2)
fatigue (Investigations) | 13 (13)
gastritis (Investigations) | 2 (2)
hyperglycemia (Investigations) | 4 (4)
HCT (Investigations) | 4 (4)
hemorrhoids (Investigations) | 2 (2)
Hyperbili (Investigations) | 6 (6)
hyperalbumin (Investigations) | 2 (2)
Hypoalbumin (Investigations) | 5 (5)
Hypokalemia (Investigations) | 3 (3)
Hypomagnesium (Investigations) | 3 (3)
hyponatremia (Investigations) | 7 (7)
infection-abdomen (Investigations) | 2 (2)
lymphopenia (Investigations) | 3 (3)
nausea (Investigations) | 5 (5)
neuropathy (Investigations) | 4 (4)
pain-abdomen (Investigations) | 5 (5)
pain-extremeties (Investigations) | 4 (4)
Pain-general/tumor (Investigations) | 8 (8)
puritis (Investigations) | 5 (5)
rash (Investigations) | 11 (11)
thrmbocytopenia (Investigations) | 12 (12)
URI (Investigations) | 3 (3)
WBC (Investigations) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No